CLINICAL TRIAL: NCT07368374
Title: THE EFFECTS OF CİTRUS AND CLOVE OİL AROMATHERAPY ON FATİGUE LEVEL, SLEEP, AND QUALİTY OF LİFE İN OLDER ADULTS
Brief Title: EFFECTS OF CİTRUS AND CLOVE OİL AROMATHERAPY İN OLDER ADULTS
Acronym: ARTICLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, İbrahim Duman, Lecturer, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ERU-SBF-ID-01
Record Dates: First submitted 2025-09-23; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Aromatherapy
Keywords: aromatherapy; citrus oil; clove oil; older adults

STUDY DESIGN:
Intervention Model Description: This research is a mixed-pattern study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Bu çalışmada çift kör tasarım uygulanacaktır. Birinci körleme, katılımcılara yöneliktir; katılımcılar hangi gruba (müdahale ya da placebo kontrol) dâhil edildiklerini bilmeyeceklerdir. İkinci körleme, ön test ve son test verilerini toplayan anketörlere (Anketör 1 ve Anketör 2) yöneliktir; bu anketörler de katılımcıların hangi grupta yer aldığını bilmeyecektir.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Citrus Oil Aromatherapy Arm, (Experimental): Older adults receiving inhalation aromatherapy with 2 drops of pure citrus oil for 2 minutes, 3 times a week, for one month (12 sessions in total).
  Interventions: Other: Intervention Group 1
- Clove Oil Aromatherapy Arm (Experimental): Older adults receiving inhalation aromatherapy with 2 drops of pure clove oil for 2 minutes, 3 times a week, for one month (12 sessions in total).
  Interventions: Other: Intervention Group 2
- Placebo Control Arm (Placebo Comparator): Older adults not receiving any aromatherapy intervention (or receiving standard care only).
  Interventions: Other: Placebo Control Group

INTERVENTIONS:
Other: Intervention Group 1 — Intervention 1 (Citrus Oil) Group: This group receives treatment 3 times a week (Mondays, Wednesdays, and Fridays between 13:00 and 14:00), for a total of 12 sessions over one month, with 2 drops of citrus oil applied to a 6x6 cm gauze pad for 2 minutes in each session.
  Arms: Citrus Oil Aromatherapy Arm,
Other: Intervention Group 2 — This group undergoes a total of 12 sessions over one month, 3 times a week (Mondays, Wednesdays, and Fridays between 13:00 and 14:00), each session involves applying 2 drops of clove oil for 2 minutes, using a 6x6 cm gauze pad in each application.
  Arms: Clove Oil Aromatherapy Arm
Other: Placebo Control Group — This group undergoes a treatment three times a week (Mondays, Wednesdays, and Fridays between 13:00 and 14:00), a total of 12 sessions over one month, and in each session, 2 drops of almond oil are applied to a 6x6 cm gauze pad for 2 minutes.
  Arms: Placebo Control Arm

SUMMARY:
This study aimed to determine the effects of citrus and clove oil aromatherapy, administered via inhalation (2 drops, 2 minutes, 3 times a week for one month), on fatigue level, sleep quality, and quality of life in older adults.

Research Hypotheses

H11: Inhalation aromatherapy with 2 drops of pure citrus oil administered for 2 minutes, 3 times a week, for a total of 12 sessions over one month is effective on fatigue level in older adults.

H01: Inhalation aromatherapy with 2 drops of pure citrus oil administered for 2 minutes, 3 times a week, for a total of 12 sessions over one month is not effective on fatigue level in older adults.

H12: Inhalation aromatherapy with 2 drops of pure citrus oil administered for 2 minutes, 3 times a week, for a total of 12 sessions over one month is effective on sleep quality in older adults.

H02: Inhalation aromatherapy with 2 drops of pure citrus oil administered for 2 minutes, 3 times a week, for a total of 12 sessions over one month is not effective on sleep quality in older adults.

H13: Inhalation aromatherapy with 2 drops of pure citrus oil administered for 2 minutes, 3 times a week, for a total of 12 sessions over one month is effective on quality of life in older adults.

H03: Inhalation aromatherapy with 2 drops of pure citrus oil administered for 2 minutes, 3 times a week, for a total of 12 sessions over one month is not effective on quality of life in older adults.

H14: Inhalation aromatherapy with 2 drops of pure clove oil administered for 2 minutes, 3 times a week, for a total of 12 sessions over one month is effective on fatigue level in older adults.

H04: Inhalation aromatherapy with 2 drops of pure clove oil administered for 2 minutes, 3 times a week, for a total of 12 sessions over one month is not effective on fatigue level in older adults.

H15: Inhalation aromatherapy with 2 drops of pure clove oil administered for 2 minutes, 3 times a week, for a total of 12 sessions over one month is effective on sleep quality in older adults.

H05: Inhalation aromatherapy with 2 drops of pure clove oil administered for 2 minutes, 3 times a week, for a total of 12 sessions over one month is not effective on sleep quality in older adults.

H16: Inhalation aromatherapy with 2 drops of pure clove oil administered for 2 minutes, 3 times a week, for a total of 12 sessions over one month is effective on quality of life in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are: • 65 years of age or older

  * Registered at the 60+ Refreshment University campus
  * Can understand and communicate in Turkish
  * Have a score of ≥24 on the Standardized Mini Mental State Examination (SMMT)
  * Have a visual similarity scale (VAS-S) score of 4 or higher for sleep problems within the past week
  * Have a visual similarity scale (VAS-F) score of 4 or higher for fatigue level within the past week
  * Have agreed to participate in the study will be included in the study.

Exclusion Criteria:

* Those with a known allergy/sensitivity to citrus or clove oil,
* Those diagnosed with any respiratory disease (asthma, COPD, etc.),
* Those with any health condition that impairs their ability to smell will not be included in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue level assessed by the Multidimensional Fatigue Inventory (MFI-20) | Baseline and at the end of the 4-week intervention period
  Fatigue level will be assessed using the Multidimensional Fatigue Inventory (MFI-20), a validated self-report questionnaire. Prior to the initiation of the aromatherapy intervention, baseline MFI-20 data will be collected through face-to-face interviews conducted by Assessor 1. Following the completion of the four-week intervention period, the MFI-20 will be re-administered through face-to-face interviews by Assessor 2. The primary outcome will be the mean change in total MFI-20 score from baseline to post-intervention. Comparisons will be conducted between the intervention groups and the placebo control group.
Change in insomnia complaints and sleep quality assessed by the Basic Insomnia and Sleep Quality Scale (BaSIQS) | Baseline and at the end of the 4-week intervention period
  Insomnia complaints and sleep quality will be assessed using the Basic Insomnia and Sleep Quality Scale (BaSIQS), a validated self-report questionnaire. Baseline measurements will be collected through face-to-face interviews conducted by Assessor 1 prior to the initiation of the aromatherapy intervention. Following the completion of the four-week intervention period, the BaSIQS will be re-administered through face-to-face interviews by Assessor 2. The primary outcome will be the mean change in total BaSIQS score from baseline to post-intervention. Comparisons will be made between the aromatherapy intervention groups and the placebo control group.

SECONDARY OUTCOMES:
Change in quality of life assessed by the Older People's Quality of Life Questionnaire-Brief (OPQOL-Brief) | Baseline and at the end of the 4-week intervention period
  Quality of life will be assessed using the Older People's Quality of Life Questionnaire-Brief (OPQOL-Brief), a validated self-report instrument. Baseline measurements will be collected through face-to-face interviews conducted by Assessor 1 prior to the initiation of the aromatherapy intervention. Following the completion of the four-week intervention period, the OPQOL-Brief will be re-administered through face-to-face interviews by Assessor 2. The primary outcome will be the mean change in total OPQOL-Brief score from baseline to post-intervention. Comparisons will be made between the aromatherapy intervention groups and the placebo control group.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD), even if anonymized, will not be shared with researchers outside the primary study team. The collected individual-level data will be used solely for the purposes of this study and will be protected in accordance with ethical approval and informed consent procedures. Study findings will be reported only in aggregate form, and no external access to individual participant data will be provided.

REFERENCES:
- See also: Related Info — https://avesis.erciyes.edu.tr/yayin/c59f5d6f-96be-4aad-83ad-4bc0c136eb31/the-effect-of-lavender-essential-oil-aromatherapy-on-anxiety-and-fatigue-in-patients-with-implantable-cardioverter-defibrillator-randomized-controlled-trial
- Available data/document: Study Protocol — https://avesis.erciyes.edu.tr/yayin/c59f5d6f-96be-4aad-83ad-4bc0c136eb31/the-effect-of-lavender-essential-oil-aromatherapy-on-anxiety-and-fatigue-in-patients-with-implantable-cardioverter-defibrillator-randomized-controlled-trial